CLINICAL TRIAL: NCT07083869
Title: Testing the Insomnia Coach Mobile App With Veterans With Insomnia and PTSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Eric Kuhn, Principal Investigator, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-79382
Record Dates: First submitted 2025-07-03; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Insomnia; Posttraumatic Stress Disorder (PTSD)
Keywords: Mobile app; Veteran; Cognitive Behavioral Therapy for Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insomnia Coach Mobile App (Experimental): Insomnia Coach is a mobile application that provides psychoeducation and self-management tools for insomnia symptoms based on cognitive behavioral therapy for insomnia (CBT-I).
  Interventions: Behavioral: Insomnia Coach
- Sleep Well Website (Active Comparator): Sleep Well is a website that is mobile enabled that provides psychoeducation about healthy sleep habits that is based on NIH Health Guide to Health Sleep and VA's Whole Health Change Your Habits to Sleep Better.
  Interventions: Behavioral: Sleep Well

INTERVENTIONS:
Behavioral: Insomnia Coach — Insomnia Coach is a mobile application that provides psychoeducation and self-management tools for insomnia symptoms based on cognitive behavioral therapy for insomnia (CBT-I)
  Arms: Insomnia Coach Mobile App
Behavioral: Sleep Well — Sleep Well is a website that is mobile enabled that provides psychoeducation about healthy sleep habits that is based on NIH Health Guide to Health Sleep and VA's Whole Health Change Your Habits to Sleep Better.
  Arms: Sleep Well Website

SUMMARY:
The objective of this randomized controlled trial of the Insomnia Coach mobile app is to evaluate the potential effects of app use on reducing insomnia symptoms among Veterans with significant insomnia and PTSD symptoms. It is also intended to evaluate the impact of the app on other outcomes, including PTSD, depression, and anxiety symptoms, and psychosocial functioning. Finally, the study is designed to assess perceptions of Insomnia Coach regarding its perceived helpfulness, satisfaction, and likes/dislikes to inform its continued improvement. The results of this study will inform the next steps of research evaluating Insomnia Coach with Veterans with significant insomnia and PTSD symptoms, namely a larger-scale, VA ORD or NIH funded randomized controlled trial.

DETAILED DESCRIPTION:
There is a high rate of insomnia among Veterans, particularly those who have been exposed to potentially traumatic situations (e.g., combat exposure) yet few of these Veterans receive cognitive-behavioral therapy for insomnia (CBT-I), a first-line treatment for insomnia. In this pilot study we seek to evaluate if Insomnia Coach is a promising tool for individuals with traumatic stress who are experiencing sleep difficulties, and therefore, demonstrate that it has the potential to address a need using a very cost-effective, widely accessible, scalable solution that would warrant more rigorous evaluation (e.g., a full-scale RCT).

Thus, in this pilot randomized controlled trial (RCT), Veterans with significant insomnia and PTSD symptoms will be recruited using hardcopy and digital flyers and 130 will be enrolled and randomized in equal numbers (1:1) to receive one of two conditions: 1) the Insomnia Coach mobile app (which is based on cognitive-behavioral therapy for Insomnia [CBT-I]) or, 2) a web-based sleep education control (i.e., Sleep Well). We will track objective use of the Insomnia Coach mobile app to assess feasibility (i.e., will participants use the app as intended). Participants will complete measures (using VA REDCap) of sleep, insomnia severity, PTSD, depression and anxiety symptoms, and functional well-being at baseline, 8 weeks (post-treatment), and 16 weeks (follow-up). At post-treatment, participants in the Insomnia Coach condition will also be asked to report their level of satisfaction with the app.

Participants will be 130 Veterans with probable insomnia and probable PTSD. Potential participants will be screened for eligibility using VA's REDCap platform. If eligible, VA REDCap will be used to administer the informed consent documents and provide participants with access to complete the baseline self-report assessments. Participants who consent and complete the baseline assessment will then be randomized with an equal probability (1:1) to conditions. Those assigned to the Insomnia Coach condition will be provided with information about how to download the research version of Insomnia Coach. Objective app use data will be monitored. Those assigned to the sleep education control will be provided with a link to access the mobile-friendly website, called "Sleep Well". No PHI/IIHI will be collected on the app (Insomnia Coach) or website (Sleep Well). Likewise, no PHI/IIHI will be disclosed via the app or website. VA REDCap will be used to administer the post-treatment assessment (at 8 weeks) and the follow-up assessment (at 16 weeks).

ELIGIBILITY:
Inclusion Criteria:

* U.S. military Veteran
* Aged 18 years or older
* Owner of smartphone or tablet with Android or iOS operating system
* Probable insomnia (i.e., ISI >=15)
* Probable PTSD (i.e., PCL-5 >=31)
* Able to read/write English
* Internet connection and active email address

Exclusion Criteria:

* Comorbid sleep disorders (apnea, RLS, narcolepsy)*
* Started or changed dosage of sleep medications or SSRIs in past 2 months
* Unstable housing
* Medical condition identifiably causing sleep problems
* Current mania or psychosis or seizure-related disorder
* Currently receiving or having recently received insomnia therapy resembling CBT-I
* Shift working
* Pregnant
* Newborn (3 mos. or younger) living in residence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI; Bastien et al., 2011) | 8 and 16 weeks
  A 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia symptoms in the past month. Items are on a scale from 0 to 4. The seven answers are added up to get a total score, with higher scores reflecting greater insomnia severity
Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 1989) | 8 and 16 weeks
  A 19-item self-report measure assessing qualities and problems associated with sleep in the past month. It generates seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. A global sleep quality score is obtained by summing the seven component scores. Higher scores reflect poorer sleep quality. The global score ranges from 0 to 21, with a cut-off score of 5 as distinguishing "good" sleepers from "poor" sleepers.
PROMIS-Sleep-Related Impairment (PROMIS-SRI; Buysse et al., 2010) | 8 and 16 weeks
  This 16-item self-report form assesses sleep-related impairment over the past seven days. Each question has five response options ranging in value from 1 to 5. To find the total raw score the values of the response to each question are summed. The raw scores are converted to a standardized T-score using conversion tables published on the PROMIS website (nihpromis.org), with higher scores indicating greater sleep/wake disturbances.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder - 7 Item (GAD-7; Spitzer et al., 2006) | 8 and 12 weeks
  This 7-item measure assesses anxiety symptom severity. Items are scored from zero to three. The whole scale score can range from 0 to 21 and cut-off scores for mild, moderate and severe anxiety symptoms are 5, 10 and 15 respectively.
Patient Health Questionnaire 8 (PHQ-8; Kroenke et al., 2009) | 8 and 16 weeks
  An 8-item self-report instrument used to assess depression severity. Since the scale is self-administered in our studies and further probing about positive responses is not feasible, the question about suicide from the PHQ-9 was removed. Items are scored 0 to 3, with the total score being the sum of the 8 items. Higher scores indicate greater depression severity, with a score of 10 or greater considered major depression, and scores of 20 or more is severe major depression.
Mobile Apps Rating Scale (MARS; Stoyanov et al., 2015) | 8 weeks
  A 20-item multidimensional, objective measure of app usability. It includes four subscales that measure an app's engagement, functionality, aesthetics, and information quality. All items are rated on a 5-point scale from "1. Inadequate" to "5. Excellent". The scores are tallied up and a mean score out of 5 is given to each of the categories scored.
System Usability Scale (SUS; Brooke, 1986) | 8 weeks
  A 10-item questionnaire of usability of products and services, including hardware, software, mobile devices, websites and applications. Items are on a 5-point scale numbered 1 to 5. Half of the items are worded negatively and half are worded positively. SUS yields a single number representing a composite measure of the overall usability of the system. To calculate the SUS score, the score contributions from each item are summed. Each item's score contribution will range from 0 to 4. For items 1,3,5,7,and 9 the score contribution is the scale position minus 1. For items 2,4,6,8 and 10, the contribution is 5 minus the scale position. Then the sum of the scores is multiplied by 2.5 to obtain the overall value of SU. SUS scores have a range of 0 to 100.
Dysfunctional Beliefs and Attitudes about Sleep (DBAS-16; Morin et al., 2007). | 8 and 12 weeks
  This 16-item self-report measures attitudes and beliefs about sleep in 4 domains: consequences of insomnia, worry and helplessness about sleep, sleep expectations, and sleep medications. Items are rated from 1 (strongly disagree) to 10 (strongly agree). An average score is calculated, with higher scores indicating stronger endorsement of unhelpful sleep cognitions.
PTSD Checklist for DSM-5 (PCL-5; Weathers et al., 2013) | 8 and 16 weeks
  A 20-item self-report questionnaire assessing PTSD symptoms in the past month. Items are on a scale from 0 to 4. The 20 item responses are summed to get a total score, with higher scores reflecting greater PTSD symptom severity
WHO QOL-BREF (Murphy et al., 2000) | 8 and 16 weeks
  This 26-item self-report measure of quality of life (QOL), life satisfaction, and personal well-being assesses the broad domains of physical health, psychological health, social relationships, and environmental factors (e.g., finances, safety). Item are rated on a variety of 1 to 5 scales with domain score items being summed to generate subscale scores with higher scores reflecting more higher QOL etc.
Fear of Sleep Inventory Short Form (FoSI-SF; Pruiksma et al., 2014) | 8 and 16 weeks
  The FoSI-SF is a 13-item self-report measure that assesses trauma-related thoughts and activities associated with sleep and the occurrence of traumas associated with the bedroom or sleep. Items are rated from 0 (not at all) to 4 (nearly every night). Total scores range from 0 to 52, with higher scores indicating greater fear of sleep.
Disturbing Dream and Nightmare Severity Index (DDNSI-15; Krakow et al., 2000) | 8 and 16 weeks
  The DDNSI is a self-report measure that assesses number of nights of nightmares, number of nightmares per week, frequency of awakenings (0 = never/rarely to 4 = always), intensity (0 = not intense to 6 = extremely severe intensity) and severity (0 = no problem to 6 = very severe problem). Scores range between 0 and 37, with a score ≥10 suggestive of nightmare disorder.

IPD SHARING:
Plan to Share IPD: No